CLINICAL TRIAL: NCT05074628
Title: Effect of Nitrofurantion Used as an Intracanal Medicament on the Intensity of Postoperative Pain and Bacterial Load Reduction Versus Calcium Hydroxide in Teeth With Necrotic Pulp: A Randomized Clinical Trial
Brief Title: Effect of Nitrofurantion Used as an Intracanal Medicament
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Mohamed Elsaber, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICM
Record Dates: First submitted 2021-10-02; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Intracanal Medication
Keywords: Nitrofurantion; necrotic pulp; Calcium Hydroxide
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Nitrofurantoin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrofurantion (Experimental): is the drug of choice for the treatment of infections caused by multidrug resistant pathogens.
  Interventions: Drug: Nitrofurantoin capsules
- Calcium Hydroxide (Active Comparator): Most commonly used intracanal medicaments . Antimicrobial activity of calcium hydroxide is related to the release of hydroxyl ions in an aqueous environment.
  Interventions: Drug: Nitrofurantoin capsules

INTERVENTIONS:
Drug: Nitrofurantoin capsules — methyl cellulose powder (MC) will be added to Nit solution to get a thick paste like consistency mixture.

SUMMARY:
The aim of this study is to clinically evaluate the effect of Nitrofurantion on Intensity of Postoperative Pain and Bacterial Load Reduction, when compared to calcium hydroxide in teeth with necrotic pulp.

DETAILED DESCRIPTION:
Nitrofurantoin has been used as a treatment for UTI since the 1950s. Evidence suggested that nitrofurantoin has excellent safety profile and lower resistance rates compared to recently introduced antimicrobials, recommending it as the first-line agent. Nitrofurantoin is convert to reactive intermediates by bacterial Nitroreductases. These intermediates were shown to attack bacterial ribosomal proteins non-specifically, causing complete inhibition of protein synthesis. In MIC, Nitrofurantoin specifically inhibit enzyme synthesis in bacteria (24). The lack of clinically significant bacterial resistance development to Nitrofurantoin is likely due to the multiple sites of attack and multiple mechanisms of action. Achievement of high local levels and low serum concentrations, and its effectiveness against both gram-negative and gram-positive bacteria provide many advantages that many of the newer agents do not have. After searching the database there is no clinical studies found yet on the effect of Nitrofurantoin antibiotic used as intracanal medicament in teeth with necrotic pulp. The aim of this study is to clinically evaluate the effect of Nitrofurantion on Intensity of Postoperative Pain and Bacterial Load Reduction, when compared to calcium hydroxide in teeth with necrotic pulp.

ELIGIBILITY:
Inclusion Criteria:

* 1- Age between 18-50 years old. 2-Males or females. 3-Healthy patients whom are categorized as I or II according to The American Society of Anesthesiologists. (ASA I or II) 4-Patients' accepting to participate in the trial. 5-Patients who can understand pain scale and can sign the informed consent. 6- Mandibular Single rooted premolars, having single root canal:

  * Diagnosed clinically with pulp necrosis.
  * Absence of spontaneous pain
  * Slight widening in the periodontal membrane space or with periapical radiolucency not exceeding 2*2 mm radiographically.
  * Normal occlusal contact with opposing teeth.

Exclusion Criteria:

* 1- Medically compromised patients having significant systemic disorders (ASA III or IV).

  2-If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively as it might alter their pain perception.

  3-Pregnant women: to avoid radiation exposure, anaesthesia, medication and hormonal Fluctuation that might increase pain prevalence.

  4-Patients reporting bruxism, clenching, TMJ problems or traumatic occlusion: to avoid further pressure on inflamed tooth which induce subsequent irritation and inflammation.

  5-Patients with two or more adjacent teeth requiring endodontic treatment. 6- Teeth that requires further procedural steps or multidisciplinary approach, which is out of this experiment's scope: i.Association with swelling or fistulous tract. ii. Acute periapical abscess. iii. Mobility Grade II or III. iv. Pocket depth more than 5mm. v. Previous root canal treatment. vi. Non-restorable. vii. Immature root. Vii. Radiographic evidence of external or internal root resorption, vertical root fracture, perforation, calcification.

  7-Inability to perceive the given instructions.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 2 Weeks
  measured using numerical rating scale (NRS), 6, 12, 24, 48 hours:

SECONDARY OUTCOMES:
Bacterial load reduction | 2 Weeks
  determined by bacterial counting using agar culture technique after root canal preparation (CFU/ml).
Incidence of inter-appointment flare up | 2 Weeks
  measured using visual analog scale of postoperative swelling (VAS).
Incidence of analgesic intake | 2 Weeks
  numerical counting.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alrahman MSA, Faraj BM, Dizaye KF. Assessment of Nitrofurantoin as an Experimental Intracanal Medicament in Endodontics. Biomed Res Int. 2020 Feb 18;2020:2128473. doi: 10.1155/2020/2128473. eCollection 2020. PMID 32149086